CLINICAL TRIAL: NCT05669313
Title: The Effects of Hypothermia and Acidosis on Coagulation During Treatment With Rivaroxaban Measured With Rotational Thromboelastometry (ROTEM)
Brief Title: The Effects of Hypothermia and Acidosis on Coagulation During Treatment With Rivaroxaban Measured With ROTEM
Status: Completed | Type: Observational
Sponsor: Thomas Kander (Other)
Responsible Party: Sponsor-Investigator, Thomas Kander, Associate Professor, Region Skane
Organization: Region Skane (Other)
Other Study IDs: Hypoth.Acidosis.Rivarox.ROTEM
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Trauma; Hypothermia; Acidosis; Bleeding
MeSH Terms: conditions — Wounds and Injuries; Hypothermia; Acidosis; Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients planned for treatment with rivaroxaban
  Interventions: Drug: Rivaroxaban 15 MG

INTERVENTIONS:
Drug: Rivaroxaban 15 MG — Rivaroxaban 15 mg after inclusion and on the morning after inclusion, i.e., before blood sampling

SUMMARY:
Rivaroxaban, a non-vitamin K oral anticoagulants, is increasingly used to prevent stroke in patients with atrium fibrillation. It has previously been demonstrated that a point-of-care coagulation instrument (ROTEM) can detect the effects of rivaroxaban. Further, the ROTEM instrument can also detect the effects of hypothermia and acidosis. Given that trauma induced coagulopathy is enhanced by both hypothermia, acidosis and rivaroxaban, the investigators want to investigate any synergistic effects between hypothermia or acidosis and rivaroxaban. In an attempt to do so the investigators designed the current experimental study with the purpose to investigate the effects of rivaroxaban together with hypothermia or acidosis using the ROTEM assay EXTEM. The hypothesis is that a synergistic prolongation of hypothermia or acidosis and rivaroxaban can be detected in the initiation of clot formation demonstrated in the primary outcome variable, clotting time of the ROTEM assay EXTEM. Secondary outcome variables include direct effect on clotting time and direct and synergistic effects on clot formation time and alfa angle of hypothermia and acidosis detected in the ROTEM assay EXTEM.

DETAILED DESCRIPTION:
Non-vitamin K oral anticoagulants (NOACs) are widely used as prophylaxis against ischaemic stroke in patients with atrial fibrillation and have replaced vitamin K antagonists (VKA) in many case. Compared to the latter they have demonstrated reduced incidence of stroke, all-cause mortality, and a reduced risk of bleeding, except for gastrointestinal bleeding. According to guidelines from the European Society of Cardiology it is recommended that patients with atrial fibrillation (AF) and adequate CHA¬2DS2-VASc score (2 for men and 3 for women) preferentially are treated with NOAC rather than VKA, except in cases with significant mitral stenosis or mechanical heart valves. Both the prevalence of patients with AF and of patients treated with NOAC have increased in the last decade.

The NOACs available in clinical practice include one thrombin inhibitor (dabigatran) and three factor Xa inhibitors (apixaban, edoxaban, rivaroxaban) [3]. These drugs drive a patient's blood further from clotting toward bleeding, and managing this tendency is important for clinicians during haemorrhage or coagulopathy, which both occur e.g., in the setting of trauma.

Trauma is a significant cause of mortality worldwide and among patients suffering from traumatic injuries the leading cause of preventable death is uncontrolled bleeding. Coagulopathy has been shown to contribute to bleeding in as many as one third of trauma cases, predicting organ failure and mortality. This trauma induced coagulopathy (TIC) is associated with hypothermia and acidosis. To prevent further coagulopathy current trauma guidelines recommend that both body temperature and pH are kept within normal reference range. Coagulopathy, hypothermia, and acidosis have collectively come to be known as the 'lethal triad'.

For trauma patients, hypothermia is associated with larger usage of blood products and increased mortality/morbidity. How hypothermia affects haemostasis and blood loss has been investigated in several studies. Hypothermia has been shown to worsen the function of secondary haemostasis through temporary reduction of fibrinogen synthesis and inhibition of the initiation phase of thrombin generation.

Hypothermia and acidosis often coexist and body temperatures of less than 35 degrees Celsius have been shown to correlate with acidosis. The effects of hypothermia and acidosis on whole blood coagulation in vitro, have previously been studied using Rotational thromboelastometry (ROTEM). For hypothermia, a significant increase in coagulation time (CT) and clot formation time (CFT) was observed, while acidosis alone did not produce these significant effects. Interestingly however, combining acidosis with hypothermia worsened the effects of the latter, providing increases in CT and CFT at higher temperatures, and a synergistic effect between acidosis and hypothermia could be demonstrated.

The ROTEM assay EXTEM has previously been shown to be more sensitive to elevated concentrations of NOAC in blood compared with other ROTEM assays, with a demonstrated linear relationship between increasing concentrations of NOAC and prolonged clotting time (CT).

In summary, the EXTEM-assay can detect the effect of rivaroxaban as well as effects of acidosis and hypothermia. However, to the best of the investigators knowledge the possibility of any synergistic effects of acidosis or hypothermia together with NOACs on the EXTEM-assay has never been explored. Given the increased prevalence of patients treated with NOAC and the importance of acidosis and hypothermia in critical bleeding the investigators designed the current experimental study with the purpose to investigate the effects of Rivaroxaban together with hypothermia or acidosis using the ROTEM assay EXTEM. The hypothesis is that a synergistic prolongation of hypothermia or acidosis and rivaroxaban can be detected in the initiation of clot formation demonstrated in the primary outcome variable, CT of the ROTEM assay EXTEM. Secondary outcome variables include direct effect on CT and direct and synergistic effects on CFT and AA of hypothermia and acidosis detected in the ROTEM assay EXTEM.

Methods Adult patients >18 years of age, reporting to the emergency department during office hours at Skåne University Hospital Lund, Sweden that are planned for rivaroxaban treatment will be included. Baseline blood samples will be taken prior to the first dose of rivaroxaban (15 mg) and a second set of blood samples will be taken at a follow up visit the next day after two doses of rivaroxaban had been taken, the later dose being taken by the patient the morning of the follow up visit and thus ensuring sampling within one half-life of rivaroxaban. On both occasions venous blood will be drawn in 2.7 ml tubes containing 0.109 M citrate (BD Vacutainer Systems, Plymouth, UK) from an antecubital vein.

At the follow up visit all patients will be asked for compliance to the rivaroxaban medication and were excluded if rivaroxaban had not been taken as prescribed. Upon the second visit a blood sample for analysis of rivaroxaban concentration wil be taken (ref. range peak value: 20 - 540 µg/L). All laboratory samples will be analysed at the accredited laboratories at Skåne University Hospital Lund or Malmö.

Immediately after blood sampling, citrate blood will be transferred to 1.5 ml plastic test tubes (Sarstedt, Micro tube 1.5 ml, Sarstedt AG & Co. KG, Nümbrecht, Germany) and divided in one temperature group and one acidosis group, each consisting of four vials.

The temperature group vials will be incubated for 20 minutes at their target goal temperatures of 28, 33, 37, and 40 degrees Celsius. The acidosis group will be incubated at 37 degrees Celsius and mixed with 15 µl of hydrochloric acid (HCl) at concentrations of 0.15 µM, 0.10 µM, 0.05 µM, or sterile water. Titration with the different concentrations of HCl will be tested prior to the current study using blood from healthy volunteers, with the goal of reaching the clinically relevant, pre-defined pH levels of 6.80, 7.00, and 7.20. After the addition of hydrochloric acid and sterile water the pH in each tube was measured using a pH-meter (Testo, Testo 230 pH/Temperature Meter, Testo SE & Co. KGaA, Lenzkirch, Germany). All tests were performed within four hours of drawing blood.

After incubation at different temperatures and the addition of HCl/sterile water, all tests will be analysed using one of two machines: the acidosis group using ROTEM using the EXTEM assay. Clotting time (CT), Alpha angle (AA), and Clot formation time (CFT) will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* any indication for starting treatment with rivaroxaban

Exclusion Criteria:

* recent medication, within the last month, with anticoagulating medication including Vitamin K antagonists and non-vitamin K antagonists, platelet inhibitors (not acetylsalicylic acid), non-steroidal anti-inflammatory drugs
* previously diagnosed coagulopathy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending the emergency department at Skåne University Hospital in Lund, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-09-04 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Clotting time of the ROTEM assay EXTEM | From inclusion to the day after inclusion when the second blood sample was taken
  Measured in seconds

SECONDARY OUTCOMES:
Clot formation time of the ROTEM assay EXTEM | From inclusion to the day after inclusion when the second blood sample was taken
  Measured in seconds
Alpha Angle of the ROTEM assay EXTEM | From inclusion to the day after inclusion when the second blood sample was taken
  Measured in degrees of the slope of the Temogram

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sunnersjo L, Ymen I, Schott U, Hillarp A, Unden J, Kander T. Synergistic effects of rivaroxaban and hypothermia or acidosis on coagulation initiation measured with ROTEM(R): a prospective observational study. Thromb J. 2024 Oct 18;22(1):91. doi: 10.1186/s12959-024-00661-0. PMID 39425155